CLINICAL TRIAL: NCT02252380
Title: A Feasibility Clinical Trial of the Magnetic Resonance Guided Focused Ultrasound (MRgFUS) for the Management of Treatment-Refractory Movement Disorders
Brief Title: ExAblate Transcranial MRgFUS for the Management of Treatment-Refractory Movement Disorders
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MD003
Record Dates: First submitted 2014-09-26; First posted 2014-09-30 (Estimated); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Movement Disorders; Essential Tremor; Holmes Tremor; Parkinson's Disease; Wilson's Disease; Huntington's Disease; Dystonia; Tardive Dyskinesia; Orofacial Dyskinesias
MeSH Terms: conditions — Movement Disorders; Essential Tremor; Ataxia; Parkinson Disease; Hepatolenticular Degeneration; Huntington Disease; Dystonia; Tardive Dyskinesia; Dyskinesias

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Transcranial ExAblate System (Experimental): Transcranial ExAblate System (MRgFUS)
  Interventions: Device: Transcranial ExAblate System

INTERVENTIONS:
Device: Transcranial ExAblate System — MR Guided Focused Ultrasound
  Other Names: MRgFUS; Focused Ultrasound; FUS

SUMMARY:
The proposed study is to evaluate the effectiveness of ExAblate Transcranial MRgFUS as a tool for creating a unilateral lesion in the Vim thalamus or the globus pallidus (GPi) in patients with treatment-refractory symptoms of movement disorders.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and initial effectiveness of MRI-guided focused ultrasound thermal ablation of a designated area in the brain of patients suffering from movement disorder symptoms:

* FUS under MRI-guidance and MRI-based thermometry can be safely delivered to patients suffering from treatment-refractory movement disorders through an intact human skull with a low risk of transient adverse effects as evaluated during follow-up of up to 12-months.
* A pre-defined target volume inside the brain can be accurately ablated, as demonstrated on post-treatment MRI.
* Lesions generated with ExAblate Neuro will result in clinical effects that are similar to those seen with ablative procedures using other surgical techniques (e.g. RF procedure).

ELIGIBILITY:
Inclusion Criteria:

* Men and women, between 18 and 85 years, inclusive.
* Subjects who are able and willing to give consent and able to attend all study visits.
* A movement disorder symptom that has been deemed treatment-refractory by a movement disorder neurologist, including:

  o akathisia, akinesia, athetosis, bradykinesia, chorea, dystonia, tremor, myoclonus, dyskinesia, spasms, tics
* Medication-refractoriness as determined by an adequate dose and duration of standard movement disorders treatment as determined by a specialist neurologist (e.g. a trial of primidone and propranolol for ET)
* Able to communicate sensations during the ExAblate Neuro treatment
* Stable doses of all medications for 30 days prior to study entry and for the duration of the study.

Exclusion Criteria:

* Patients with unstable cardiac status including:

  * Unstable angina pectoris on medication
  * Patients with documented myocardial infarction within six months of protocol entry
  * Congestive heart failure requiring medication (other than diuretic)
  * Patients on anti-arrhythmic drugs
* Severe hypertension (diastolic BP > 100 on medication)
* Patients with standard contraindications for MR imaging such as non-MRI compatible implanted metallic devices including cardiac pacemakers, size limitations, etc.
* History of abnormal bleeding and/or coagulopathy (including deep venous thrombosis)
* Cerebrovascular disease (multiple CVA or CVA within 6 months)
* Symptoms and signs of increased intracranial pressure (e.g. headache, nausea, vomiting, lethargy, and papilledema)
* Untreated, uncontrolled sleep apnea
* Active or suspected acute or chronic uncontrolled infection
* History of intracranial hemorrhage
* Individuals who are not able or willing to tolerate the required prolonged stationary supine position during treatment
* Are participating or have participated in another clinical trial in the last 30 days
* Patients unable to communicate with the investigator and staff.
* Presence of any other neurodegenerative disease like multisystem atrophy, progressive supranuclear palsy, dementia with Lewy bodies, and Alzheimer's disease.
* Patients with a history of seizures within the past year
* Patients with psychiatric illness that are not well controlled. Any presence of psychosis will be excluded.
* Patients with risk factors for intraoperative or postoperative bleeding (platelet count less than 100,000 per cubic millimeter) or a documented coagulopathy
* Patients with brain tumors
* Any illness that in the investigator's opinion preclude participation in this study.
* Pregnancy or lactation.
* Patient is unable to provide his own consent for any reason.
* Legal incapacity or limited legal capacity.
* Patients who have DBS or a prior stereotactic ablation of the basal ganglia
* History of immunocompromise, including patient who is HIV positive
* Known life-threatening systemic disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-05; Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Severity of Device and Procedure Related Complications | At the time of ExAblate procedure
  Safety will be evaluated individually for each subject who is treated

CONTACTS AND LOCATIONS:
Overall Officials: Andres Lozano, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (2):
- Canada (2):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Germann J, Santyr B, Boutet A, Sarica C, Chow CT, Elias GJB, Vetkas A, Yang A, Hodaie M, Fasano A, Kalia SK, Schwartz ML, Lozano AM. Comparative neural correlates of DBS and MRgFUS lesioning for tremor control in essential tremor. J Neurol Neurosurg Psychiatry. 2024 Jan 11;95(2):180-183. doi: 10.1136/jnnp-2022-330795. PMID 37722831
- [Derived] Yamamoto K, Sarica C, Elias GJB, Boutet A, Germann J, Loh A, Joel SE, Bigioni L, Gwun D, Gramer R, Li SX, Zemmar A, Vetkas A, Algarni M, Devenyi G, Chakravarty M, Hynynen K, Scantlebury N, Schwartz ML, Lozano AM, Fasano A. Ipsilateral and axial tremor response to focused ultrasound thalamotomy for essential tremor: clinical outcomes and probabilistic mapping. J Neurol Neurosurg Psychiatry. 2022 Aug 22:jnnp-2021-328459. doi: 10.1136/jnnp-2021-328459. Online ahead of print. PMID 35995551
- [Derived] Kapadia AN, Elias GJB, Boutet A, Germann J, Pancholi A, Chu P, Zhong J, Fasano A, Munhoz R, Chow C, Kucharczyk W, Schwartz ML, Hodaie M, Lozano AM. Multimodal MRI for MRgFUS in essential tremor: post-treatment radiological markers of clinical outcome. J Neurol Neurosurg Psychiatry. 2020 Sep;91(9):921-927. doi: 10.1136/jnnp-2020-322745. Epub 2020 Jul 10. PMID 32651242
- [Derived] Fasano A, Llinas M, Munhoz RP, Hlasny E, Kucharczyk W, Lozano AM. MRI-guided focused ultrasound thalamotomy in non-ET tremor syndromes. Neurology. 2017 Aug 22;89(8):771-775. doi: 10.1212/WNL.0000000000004268. Epub 2017 Jul 26. PMID 28747452